CLINICAL TRIAL: NCT01166165
Title: Effect of Cholecalciferol on 24-hr ABPM and Vasoactive Hormones in Patients With Hypertension.
Brief Title: Effect of Vitamin D Replacement During Winter Months in Patients With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, DMSci, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBP-TL-2010-2; M-20100120 (Other: The Regional Committee on Biomedical Research Ethics)
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension; Vitamin D Deficiency
Keywords: Hypertension; blood pressure; vitamin d; winter; cholecalciferol; arterial stiffness; renin; angiotensin; aldosterone; calcium
MeSH Terms: conditions — Hypertension; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Active Comparator)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — 3 tablets of 1000 IU daily for 20 weeks
  Arms: Cholecalciferol
Drug: Placebo — 3 placebo tablets daily for 20 weeks
  Arms: Placebo

SUMMARY:
High blood pressure is related to increased risk of cardiovascular disease and death, and accounts for approximately 8 mill deaths worldwide each year. Blood pressure exhibits a seasonal variation with a tendency to increase during winter months. Vitamin D deficiency is more common during months where UVB radiation from the sun is absent, and vitamin D has been associated with high blood pressure. This study will evaluate the effect of vitamin D replacement during winter months on blood pressure and vasoactive hormones in patients with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Well-regulated arterial hypertension
* Office blood pressure > 120/70 mmHg

Exclusion Criteria:

* Pregnancy or nursing
* Cancer
* Alcohol abuse
* Continuous glucocorticoid or NSAID treatment
* 24-hour blood pressure > 150/95 mmHg
* Hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
24-hour systolic blood pressure | 20 weeks

SECONDARY OUTCOMES:
Plasma renin concentration | 20 weeks
Plasma concentration of angiotensin II | 20 weeks
Plasma concentration of aldosterone | 20 weeks
Plasma concentration of c-reactive protein | 20 weeks
Urine albumin creatinine ratio | 20 weeks
Urine calcium creatinine ratio | 20 weeks
Plasma concentration of 25-hydroxycholecalciferol | 5 weeks
Serum concentration of FGF-23 | 20 weeks
Augmentation index and central blood pressure | 20 weeks
Pulse wave velocity | 20 weeks
Heart rate variability | 20 weeks
Plasma concentration of ionized calcium | 5 weeks
Plasma concentration of phosphate | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Larsen, M.D., Principal Investigator — Departments of Medical Research, Holstebro Hospital
Locations (1):
- Department of Medical Research, Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Larsen T, Mose FH, Bech JN, Hansen AB, Pedersen EB. Effect of cholecalciferol supplementation during winter months in patients with hypertension: a randomized, placebo-controlled trial. Am J Hypertens. 2012 Nov;25(11):1215-22. doi: 10.1038/ajh.2012.111. Epub 2012 Aug 2. PMID 22854639